CLINICAL TRIAL: NCT07183488
Title: Metabolic Effects of Short-Chain Fatty Acids in Healthy Individuals
Acronym: SCFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-25038908
Record Dates: First submitted 2025-08-27; First posted 2025-09-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healhty; Other: Short-Chain Fatty Acid (SCFA); Other: Butyrate (C4); Other: Propionate (C3)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Female (Experimental)
  Interventions: Other: Propionate followed by Butyrate; Other: Butyrate followed by Propionate
- Male (Experimental)
  Interventions: Other: Propionate followed by Butyrate; Other: Butyrate followed by Propionate

INTERVENTIONS:
Other: Propionate followed by Butyrate — The participants will consume Short-chain fatty acid propionate (SCFA-PRO) followed by Short-Chain Fatty Acid Butyrate (SCFA-BUT).
  Arms: Male
Other: Butyrate followed by Propionate — • The participants will consume Short-chain fatty acid Butyrate (SCFA-BUT) followed by Short-Chain Fatty Acid Propionate (SCFA-PRO).
  Arms: Male
Other: Propionate followed by Butyrate — • The participants will consume Short-Chain Fatty Acid propionate (SCFA-PRO) followed by Short-Chain Fatty Acid Butyrate (SCFA-BUT).
  Arms: Female
Other: Butyrate followed by Propionate — The participants will consume Short-Chain Fatty Acid Butyrate (SCFA-BUT) followed by Short-Chain Fatty Acid Propionate (SCFA-PRO).
  Arms: Female

SUMMARY:
The primary objective of this study is to investigate the acute physiological and metabolic effects of ingesting the short-chain fatty acids (SCFA)s propionate (three carbon atoms long; C3:0) and butyrate (C4:0) in healthy men and women. This aim will be addressed through a block-randomized cross-over study including two visits with acute intake of propionate and butyrate, respectively.

The hypothesis is that plasma ketone body levels will increase during the first three hours after intake of butyrate, but not propionate, in healthy individuals in the overnight fasted state.

DETAILED DESCRIPTION:
The study will be conducted as a block-randomized cross-over study in healty participants (n=10). The participants will undergo two experimental days of three hours separated by a two to four weeks wash-out period. At the test days, participants will consume 3 grams of either propionate or butyrate in the form of sodium-propionate or sodium-butyrate together with 250 ml of water. The order of ingestion is determined by randomization.

The day prior to the experimental days, participants will consume a standardized control dinner and evening snack and abstain from alcohol and vigorous physical activity to ensure similar conditions on the experimental days. The standardized meal will be provided to the participants. On the test days, participants will be instructed to arrive by passive transport in an overnight fasted state (10 hours). Upon arrival, a DXA scan will be performed, after which a catheter will be inserted into an antecubital vein. Following 30 minutes of supine rest, baseline measurements will be performed, including indirect calorimetry, blood pressure measurement, flow-mediated vasodilation (FMD), and a fasting venous blood sample. Participants will then ingest 3 grams of propionate or butyrate within 5 minutes, together with 250 ml of water. After ingestion, participants will remain resting in bed for 3 hours, during which blood samples (15 ml each) will be collected continuously throughout the test day. Indirect calorimetry, blood pressure measurements, and FMD will be repeated at various time points post-ingestion. The test day will end with an ad libitum meal. The entire procedure will be repeated on the second test day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age between 18-40 years old
* BMI between 18.5-29

Exclusion Criteria:

* Diabetes
* Kidney- or liver disease
* Pregnant, lactating or planning to become pregnant within the study period
* Supplementation with SCFAs
* Supplementation with B12 vitamin
* Special dietary habits (e.g. vegan/ketogenic diet)
* Ongoing cancer treatment
* Metabolic or absorptive disorders, gastric bypass operation, or use of medication affecting metabolism or food absorption
* Crohn's disease, ulcerative colitis or short bowel syndrome
* Inability, physically or mentally, to comply with the procedure required by the study protocol as evaluated by the primary investigator, study manager or clinical responsible

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Ketone Bodies | On day 1 (test day 1) and day 2 (test day 2) at baseline (-30 min and 0 min) and post intake (10 min, 15 min, 22.5 min, 30 min, 45 min, 60 min, 90 min, 120 min, and 180 min).
  To measure the effect of Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on circulating ketone body concentrations.

SECONDARY OUTCOMES:
Glucose | On day 1 (test day 1) and day 2 (test day 2) at baseline (-30 min and 0 min) and post intake (10 min, 15 min, 22.5 min, 30 min, 45 min, 60 min, 90 min, 120 min, and 180 min).
  To measure the effect of Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on circulating glucose.
Fatty acids | On day 1 (test day 1) and day 2 (test day 2) at baseline (-30 min and 0 min) and post intake (10 min, 15 min, 22.5 min, 30 min, 45 min, 60 min, 90 min, 120 min, and 180 min).
  To measure the effect of Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on circulating Short-Chain Fatty Acids.
Flow mediated dilation measurement | On day 1 (test day 1) and day 2 (test day 2) at baseline (min -15) and post intake (min 90).
  To measure the vasodilatory effects of the short-chain fatty acids butyrate (SCFA-BUT) and propionate (SCFA-PRO) during flow-mediated dilation measurement.
Resting metabolic rate | On day 1 (test day 1) and day 2 (test day 2) at baseline (min -15) and post intake (30 min, 60 min, 120 min)
  To measure the effect of Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on resting metabolic rate.
Respiratory exchange ratio | On day 1 (test day 1) and day 2 (test day 2) at baseline (min -15) and post intake (30 min, 60 min, 120 min)
  To measure the effect of Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on respiratory exchange ratio.
Fatty Acid Composition | On day 1 (test day 1) and day 2 (test day 2) at baseline (-30 min and 0 min) and post intake (10 min, 15 min, 22.5 min, 30 min, 45 min, 60 min, 90 min, 120 min, and 180 min).
  To measure the effect of Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on fatty acid composition.
Metabolites | On day 1 (test day 1) and day 2 (test day 2) at baseline (-30 min and 0 min) and post intake (10 min, 15 min, 22.5 min, 30 min, 45 min, 60 min, 90 min, 120 min, and 180 min).
  To measure the effect of Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on circulating ketone body concentrations.
Hepatokines | On day 1 (test day 1) and day 2 (test day 2) at baseline (-30 min and 0 min) and post intake (10 min, 15 min, 22.5 min, 30 min, 45 min, 60 min, 90 min, 120 min, and 180 min).
  To measure the effect Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on circulating hepatokine concentrations.
HOMA-Index | On day 1 (test day 1) and day 2 (test day 2) at baseline (-30 min and 0 min) and post intake (10 min, 15 min, 22.5 min, 30 min, 45 min, 60 min, 90 min, 120 min, and 180 min).
  To measure the effect of Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on HOMO-index.
Satiety | On day 1 (test day 1) and day 2 (test day 2) at baseline (-15 min) and post intake (30 min, 60 min, 90 min and 120 min).
  To measure the effect of Short-Chain Fatty Acid Butyrate (SCFA-BUT) and Short-Chain Fatty Acid Propionate (SCFA-PRO) on satiety using the Visual Analog Scale (VAS), going from 0 (none) to 10 (worst possible) at a 10cm scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Copenhagen N, Denmark

IPD SHARING:
Plan to Share IPD: No